CLINICAL TRIAL: NCT03800160
Title: Greater China Metabolic and Bariatric Surgery Database
Status: Enrolling by invitation | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other); Beijing Hospital (Other Government); Peking Union Medical College Hospital (Other); Shanxi Dayi Hospital (Other); The Second Hospital of Hebei Medical University (Other); Tianjin Medical University General Hospital (Other); Inner Mongolia People's Hospital (Other); Henan Provincial People's Hospital (Other); Qilu Hospital of Shandong University (Other); The First Hospital of Hebei Medical University (Other); The Second People's Hospital of Xinxiang Henan (Unknown); Tangshan Gongren Hospital (Other); Tianjin Nankai Hospital (Other); Tianjin First Central Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Director of general surgery, principal investigator, Beijing Friendship Hospital
Other Study IDs: GC-MBD
Record Dates: First submitted 2018-05-14; First posted 2019-01-11 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Metabolic Surgery
Keywords: metabolic surgery; metabolic disease; multicenter
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Metabolic surgery, as a recognition treatment option for patients with clinical morbid obesity, is gaining increasing appreciation. In addition to substantial weight loss, emerging studies have highlighted that metabolic surgery can substantially ameliorate obesity-related metabolic diseases, including but not limited to type 2 diabetes mellitus (T2DM), hypertension, dyslipidemia, obstructive sleep apnea-hypopnea syndrome (OSAHS) and polycystic ovary syndrome (PCOS)in severely obese patients. However, further investigations with larger sample size and longer observation time still needed to clarity the efficacy and safety of metabolic surgery in Chinese patients with obesity and encouraging future research in this field.

ELIGIBILITY:
Inclusion Criteria:

* be able to receive metabolic surgery, including but not limit to LSG and LRYGB

Exclusion Criteria:

* can not be able to understand and willing to participate in this registry with signature

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with morbid obesity who are suitable and willing to accept metabolic surgical procedure and also agree with the registry
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
the excess weight loss effect of different metabolic surgeries after 1year | 1 year after surgery
  Percent excess weight loss (%EWL), %EWL=[(initial weight)-(post-op weight)]/[(initial weight)-(ideal weight)] (in which "ideal weight" is defined by the weight corresponding to a BMI of 25 kg/m2)

SECONDARY OUTCOMES:
the adverse events rate of different metabolic surgeries | 30 days after surgery
  show the surgical safety by 30 days follow-up according to guideline（such as: bleeding, leak, obstruction, re-operation for complication）
the excess weight loss effect of metabolic surgery with long-time follow-ups | 3 years
  Percent excess weight loss (%EWL), %EWL=[(initial weight)-(post-op weight)]/[(initial weight)-(ideal weight)] (in which "ideal weight" is defined by the weight corresponding to a BMI of 25 kg/m2)
the excess weight loss effect of metabolic surgery with long-time follow-ups | 5 years
  Percent excess weight loss (%EWL), %EWL=[(initial weight)-(post-op weight)]/[(initial weight)-(ideal weight)] (in which "ideal weight" is defined by the weight corresponding to a BMI of 25 kg/m2)
the excess weight loss effect of metabolic surgery with long-time follow-ups | 10 years
  Percent excess weight loss (%EWL), %EWL=[(initial weight)-(post-op weight)]/[(initial weight)-(ideal weight)] (in which "ideal weight" is defined by the weight corresponding to a BMI of 25 kg/m2)
the glycemic control level of metabolic surgery with long-time follow-ups | 1 year after surgery
  the change of HbA1c, glucose level, C-peptide and insulin levels
the glycemic control level of metabolic surgery with long-time follow-ups | 3 year after surgery
  the change of HbA1c, glucose level, C-peptide and insulin levels
the glycemic control level of metabolic surgery with long-time follow-ups | 5 year after surgery
  the change of HbA1c, glucose level, C-peptide and insulin levels
the glycemic control level of metabolic surgery with long-time follow-ups | 10 year after surgery
  the change of HbA1c, glucose level, C-peptide and insulin levels

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China